CLINICAL TRIAL: NCT03542318
Title: Effects of a Pulmonary Rehabilitation Programme on Functional and Health Status Measures in Patients With Pulmonary Fibrosis
Brief Title: Effects of Pulmonary Rehabilitation on Functional and Health Status Measures in Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Anabel Sciriha, Principal Investigator, University of Malta
Other Study IDs: 191/2011
Record Dates: First submitted 2018-05-06; First posted 2018-05-31 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Fibrosis
Keywords: Pulmonary Rehabilitation; Functional outcomes; Health Status; Exercise
MeSH Terms: conditions — Pulmonary Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active group (Experimental): Total of 60 patients were enrolled. All patients were referred for PR from the outpatient clinics of the local general hospital. Pulmonary fibrosis was confirmed through a high resonance computed tomography scan and pulmonary function testing. Participants who required modifications to their drug therapy due to exacerbations were excluded from the study. Each participant was classified according to the modified Medical Research Council dyspnoea scale
  Interventions: Other: Pulmonary Rehabilitation
- Inactive control group: A total of 60 patients were enrolled in a control group. All were referred for PR from the outpatient clinics of the local general hospital. In this group patients who requested not to carry out the intervention but participate in the investigations were enrolled. Each participant was classified according to the modified Medical Research Council dyspnoea scale, and placed in one of 5 categories (0 to 4) according to self-perceived breathlessness during daily activities

INTERVENTIONS:
Other: Pulmonary Rehabilitation — A multidisciplinary PR programme was delivered twice weekly for 12 weeks. Each class was of 2 hours in duration. The first hour had an exercise component. Inspiratory muscle training was carried out using the Respironics IMT Threshold trainer® during the class. Educational sessions covered various aspects of pulmonary fibrosis care and self-management delivered. Patients also received an individualized home exercise programme consisting of exercise similar to what was being carried out during the classes. Each participant was encouraged to perform at least 20 minutes of these exercises per day.
  Groups: Active group (Experimental)

SUMMARY:
The inclusion of Pulmonary Rehabilitation (PR) as part of the management of pulmonary fibrosis although being highly recommended and recommended in guidelines still sees studies exploring the outcomes from such an intervention limited. The present study aims to contribute to the available literature by investigating the effects of a high intensity, 12week PR programme on functional and quality of life measures in patients with a diagnosis of pulmonary fibrosis.

DETAILED DESCRIPTION:
The inclusion of Pulmonary Rehabilitation (PR) as part of the management of pulmonary fibrosis although being highly recommended and recommended in guidelines still sees studies exploring the outcomes from such an intervention limited. The present study aims to contribute to the available literature by investigating the effects of a high intensity, 12week PR programme on functional and quality of life measures in patients with a diagnosis of pulmonary fibrosis. This study reports outcomes of an observational, quasi experimental type of study. A total of 120 participants were recruited: 60 patients formed part of the active group, another 60 patients were enrolled in an inactive group. Each participant was classified according to the modified Medical Research Council dyspnoea scale and placed in one of 5 categories (0 to 4) according to self-perceived breathlessness during daily activities. The following outcomes were measured: Lung function tests including plethysmography and diffusion capacity of carbon monoxide (DLCO), functional tests (6-minute walking test, Dyspnoea Borg Scale) and Health status measures (St George's Respiratory Questionnaire and HAD score).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Pulmonary Fibrosis
* Patients had to be medically stable to participate in such a programme

Exclusion Criteria:

* Any orthopaedic or neurological condition affecting mobility
* If they required oxygen therapy this had to be used

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 120 patients were enrolled: 60 patients formed part of the active group (30 male and 30 female), another 60 patients were enrolled in an inactive, control group, 32 of which were male and 28 female participants.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | The 6MWD shall be measures at baseline and on completion of the programme at 12weeks
  The six-minute walking distance test (6MWD) was performed according to the American Thoracic Society guidelines (ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories 2002). Each patient was instructed to walk as rapidly as possible in a 30-meter corridor for the time of this test. The test was repeated twice with an interval of 30 minutes. The longest distance on a 6MWT and oxygen saturation were utilized to measure exercise capacity. Dyspnoea was scored using the Borg Category Ratio Scale (Borg 1982) measuring dyspnoea symptoms before and after the test.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression score | This outcome shall be measured at baseline and on completion of the PR programme at 12weeks
  The HAD scale was specifically developed for recognition of anxiety and depression in patients with somatic conditions. It is a validated tool which explores the symptom severity in patient with chronic diseases who have anxiety and depressive related signs. The HAD scale is divided into an anxiety (HADS-A) and a depression subscale (HADS-D) both of which contain seven items, rated 0-3, with the highest possible score for both domains being that of 21. Scores less than 8 indicate no clinical distress; scores between 8 to 10 indicate possible psychiatric morbidity and scores of 11 or more indicate pathologic levels of distress.
St George's Respiratory Questionnaire | This outcome shall be measured at baseline and on completion of the PR programme at 12weeks
  The SGRQ is a widely used questionnaire to assess health related quality of life, due to its specificity to respiratory diseases. This questionnaire consists of 50 items, separated into three domains: symptoms, activity and impact domains. Scores range from 0 to l00 for the three subscales with a summary total score. Higher scores indicate worse health status; 0 indicates no impairment and 100 indicates maximal impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Anabel Sciriha, Ph.D, Principal Investigator — Physiotherapy Department, Faculty of Health Sciences, University of Malta
Locations (1):
- Faculty of Health Sciences, Physiotherapy Department, Multiple Locations, Malta

IPD SHARING:
Plan to Share IPD: No